CLINICAL TRIAL: NCT04509063
Title: Investigating Public Enthusiasm for Mammography Screening in Denmark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-051-000001, 1835
Record Dates: First submitted 2020-06-29; First posted 2020-08-11 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Breast Neoplasm Female; Mammography Screening; Decision Making; Information Seeking Behavior
Keywords: Breast cancer; Mammography screening; Decision Making; Information Seeking Behavior
MeSH Terms: conditions — Information Seeking Behavior; Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Self administered questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Detailed information about screening harms (Other)
  Interventions: Behavioral: Information about hypothetical mammography screening without benefits
- Non-detailed information about screening harms (Other)
  Interventions: Behavioral: Information about hypothetical mammography screening without benefits

INTERVENTIONS:
Behavioral: Information about hypothetical mammography screening without benefits — We will present an online questionnaire with two types of information on the harms of screening. Then we will compare the prevalence of irrational decisions in the two arms.

SUMMARY:
Based on an American study by Scherer et al., it is hypothesized that some women will make irrational choices regarding their participation in mammography screening. Therefore, the aim is to estimate the prevalence of Danish women having an irrational preference for mammography screening even when it confers no benefits, but only harms.

DETAILED DESCRIPTION:
The prevalence of women making an irrational decision will be compared to the participation rate in the Danish screening program. The study population will consist of a random sample of women aged 44-49. Similar to the American study, two types of information will be compared (detailed vs. non-detailed information about the harms of screening). Participants will be randomised to one of two information groups. Based on the American study, it is assumed that the willingness to participate in the hypothetical screening program will be 40 percent. To achieve the desired precision in this study, a standard error of 2.5 percent is required corresponding to a confidence interval spanning approximately 35-45 percent. This will require 384 women in each group, corresponding to a total study population of 768. The survey will be sent electronically (using "e-Boks") with a link to access the online survey trial. The survey will consist of screening and cancer related questions as well as questions on age, education, and health literacy. Five questions on appraisal of health information from the Health Literacy Questionnaire will also be included. After the data collection, data will be linked to data on income, residence, civil status, education, breast cancer diagnosis, and information on whether a participant is immigrant, descendent or of Danish origin.

The original plan for the main analysis was to compare the two groups of women randomized to different information groups (detailed vs. non-detailed information about the harms of screening). However, due to lower participation rate and therefore smaller sample size than expected, information group was disregarded in the main analysis. The two groups will still be compared in a secondary analysis. This decision was made before getting access to data from the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Residence: Central Denmark Region

Exclusion Criteria:

-

Ages: 44 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 768 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Irrational preference | The outcome is assessed when women answer the questionnaire which is sent out at the same time to all women. The invited women will have 2 months to answer the questionnaire (it should only take around 15 minutes to answer). Planned from November 2020.
  Willingness to participate in mammography screening with no benefits on morbidity or mortality, only harms. Investigated by sending out questionnaire once to all women.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Not allowed by authorities.

REFERENCES:
- [Background] Scherer LD, Valentine KD, Patel N, Baker SG, Fagerlin A. A bias for action in cancer screening? J Exp Psychol Appl. 2019 Jun;25(2):149-161. doi: 10.1037/xap0000177. Epub 2018 Jul 19. PMID 30024212
- [Derived] Rossell EL, Bo A, Gronborg TK, Kristiansen IS, Borgquist S, Scherer LD, Stovring H. Danish Women Want to Participate in a Hypothetical Breast Cancer Screening with Harms and No Reduction in Mortality: A Cross-Sectional Survey. Med Decis Making. 2023 May;43(4):403-416. doi: 10.1177/0272989X231152830. Epub 2023 Feb 3. PMID 36734154

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT04509063/SAP_000.pdf